CLINICAL TRIAL: NCT07407712
Title: Better Outcomes Through Optimal Sleep in Surgical Training
Acronym: BOOST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: STH23585; 362885 (Other: IRAS)
Record Dates: First submitted 2025-12-18; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Staff

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): All participants will have a sleep intervention
  Interventions: Behavioral: Sleep intervention

INTERVENTIONS:
Behavioral: Sleep intervention — Participants will have a face-to-face consultation with a sleep consultant, which will be tailored to the specific sleep profile.
  * The consultation will include advice on sleep hygiene and may involve identifying potential sleep disorders.
  * They may be referred for additional testing at a local sleep lab if a sleep disorder is suspected.
  * If indicated by the sleep profile, they may receive short-form cognitive behavioural therapy for insomnia (CBTi), which typically involves a series of structured sessions.

SUMMARY:
This research project is investigating the impact of sleep quality on cognitive and laparoscopic surgical performance. The background to this study is the growing recognition that factors beyond technical skill, such as sleep, can significantly influence a surgeon's performance. The aim is to understand how sleep patterns affect surgeons' ability to perform surgical tasks, both technically and cognitively. After this, we will aim to see if a targeted sleep intervention has a positive impact on technical skills and cognitive performance. This is a preliminary feasibility study and is part of ongoing research by the research team.

ELIGIBILITY:
Inclusion Criteria:

* The study will recruit general surgical trainees and consultant surgeons from the Yorkshire and Humber region.
* Individuals must be willing and able to give informed consent to take part in the study.

Exclusion Criteria:

* • Participants with a previously diagnosed sleep disorder

  * Anyone who is unable to give informed consent will be excluded.
  * Individuals who are not general surgical trainees or consultant will be excluded.
  * Participants who are unable to wear the Actigraphy device continuously for two weeks, complete the daily sleep diary, or attend the in-person assessments will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in objective sleep quality as measured by Actigraphy data | From baseline to 8 weeks
  Total sleep time
Change in objective sleep quality as measured by Actigraphy data | From baseline to 8 weeks
  sleep efficiency

SECONDARY OUTCOMES:
Change in subjective sleep quality | From baseline to 8 weeks
  PSQI
Change in subjective cognitive load | From baseline to 8 weeks
  SurgTLX
Change in objective cognitive load | From baseline to 8 weeks
  HRV
Change in technical surgical performance | From baseline to 8 weeks
  GOALS framework

CONTACTS AND LOCATIONS:
Locations (1):
- Sheffield Teaching Hospitals, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No